CLINICAL TRIAL: NCT03181958
Title: Nasal High Frequency Oscillation Ventilation(NHFOV) vs. Nasal Continuous Positive Airway Pressure(NCPAP) vs Nasal Intermittent Positive Pressure Ventilation（NIPPV） as Post-extubation Respiratory Support in Preterm Infants With Respiratory Distress Syndrome:a Multicenter Randomized Controlled Trial
Brief Title: A Trial Comparing Noninvasive Ventilation Strategies in Preterm Infants Following Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other); Jiulongpo No.1 People's Hospital (Other); Chongqing Maternal and Child Health Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Peking University Third Hospital (Other); First Hospital of Tsinghua University (Other); Women and Children's Hospital, Branch of Chongqing Sanxia Central Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Quanzhou Children's Hospital (Other); Xiamen Maternity & Child Care Hospital (Other); Zhujiang Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Guangdong Academy of Medical Science and General Hospital (Other); Guangdong Women and Children Hospital (Other); Women and Children's Health Hospital of Yulin (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guiyang Maternal and Child Health Care Hospital (Other); Zunyi First People's Hospital (Industry); Lanzhou University Second Hospital (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); LanZhou University (Other); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Zhengzhou Children's Hospital, China (Other); Third Affiliated Hospital of Zhengzhou University (Other); the Maternal and Child Health Hospital of Hainan Province (Other); Bethune International Peace Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Children's Hospital of Nanjing Medical University (Other); The First Hospital of Jilin University (Other); Children's Hospital of Fudan University (Other); Maternal and Children's Healthcare Hospital of Taian (Other); The Second Hospital of Shandong University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Chengdu Women and Children's Center Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Affiliated Hospital of Southwest Medical University (Other); Shenzhen People's Hospital, The Second Medical College of Jinan University (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Kunming Children's Hospital (Other); The First People's Hospital of Yunnan (Other); First Affiliated Hospital of Kunming Medical University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Women and Children's Health Hospital of Qujing (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); The First People's Hospital of Yinchuan (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Beijing 302 Hospital (Other); Hunan Children's Hospital (Other Government); Women and Children Hospital of Qinghai Province (Other); Jiangxi Province Children's Hospital (Other); Inner Mongolia People's Hospital (Other); Mianyang Central Hospital (Other); People's Liberation Army No.202 Hospital (Other); Ningbo Women & Children's Hospital (Other); Shanghai Children's Medical Center (Other); First Affiliated Hospital of Guangxi Medical University (Other); Nanjing Medical University (Other); Qinhuangdao Maternal and Child Health Care Hospital (Other); Xuzhou Children Hospital (Other); Catholic University of the Sacred Heart (Other); The First Affiliated Hospital of Zhengzhou University (Other); Xianyang Children's Hospital (Other)
Responsible Party: Principal Investigator, Ma Juan, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201721
Record Dates: First submitted 2017-05-28; First posted 2017-06-09 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Intubated Infants Were Intend to Extubation Using Noninvasive Ventilation Strategies
Keywords: nasal high frequency oscillation ventilation(NHFOV); nasal continuous positive airway pressure(NCPAP); nasal intermittent positive pressure ventilation（NIPPV）; neonatal respiratory distress syndrome(NRDS); preterm infants
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: When the neonate had fulfilled the extubation criteria, extubation will took place with a gentle intratracheal suction. Upper airways will then be suctioned and intervention will be started immediately as follows:
  Ventilators
  * CPAP: CPAP will be provided by either variable flow or continuous flow devices, as there is no evidence that one type of CPAP generator would be better than any other.
  * NIPPV: NIPPV will be provided by any type of neonatal ventilator. Synchronization will not be applied, as many currently marketed neonatal ventilators usually do not provide it for NIPPV.
  * NHFOV: NHFOV will only be provided with piston/membrane oscillators able to provide a real oscillatory pressure with active expiratory phase (that is, Acutronic FABIAN-III, SLE 5000, Loweinstein Med LEONI+, Sensormedics 3100A). Other machines providing high frequency ventilations will not be used.
  Importantly, the randomization should be done within one hour from the extubation to avoid bias.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding towards the caregivers is impossible and blinding towards the patients makes no sense. However, outcomes' assessors will be blinded, as endpoints will be recorded by investigators not involved in patients' care. An assessor per each participating NICU will be nominated. Moreover, investigators performing the final statistical analyses will be blinded to the treatment allocation, as data collected by assessors will be inserted in the dedicated website and the arms' allocation will be re-coded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NHFOV (Experimental): neonates assigned to NHFOV will be started with the following boundaries:
  a) Paw of 10 cmH2O (can be changed in steps of 1 cmH2O within the range range 5- 16cmH2O); Paw will be titrated (within the range) according to open lung strategy, performing alveolar recruitment, similar to what is done in endotracheal high frequency oscillatory ventilation targeting a FiO2≤25-30%. Maximal allowed FiO2 will be 0.40 and SpO2 targets will be 90%-95%. b) frequency of 10Hz(can be changed in steps of 1Hz within the range 8-12Hz). c)Inspiratory time 50% (1:1).d)amplitude 25 cmH2O(can be changed in steps of 5 cmH2O within the range 25-50 cmH2o; amplitude will be titrated according to PaCO2.
  Interventions: Device: NHFOV
- NCPAP (Active Comparator): Neonates assigned to the CPAP group were initiated on a pressure of 5 cmH2O. CPAP can be raised in steps of 1 cmH2O up to 8 cmH2O. If this is not enough to maintain SpO2 between 90% and 95%, FiO2 will be added up to 0.40.
  Interventions: Device: NCPAP
- NIPPV (Experimental): neonates assigned to the NIPPV group will be started with the following parameters: a) positive end-expiratory pressure (PEEP) of 4 cmH2O (can be raised in steps of 1 cmH2O to max 8 cmH2O, according to the oxygenation).b)Peak Inspiratory Pressure (PIP) of 15 cmH2O (can be raised in steps of 1 cmH2O to max 25 cmH2O, according to oxygenation,PaCO2 levels and the chest expansion); maximal allowed FiO2 will be 0.40 and SpO2 targets will be 90-95%. c) inspiratory time (IT) will be 0.45 - 0.5 sec(according to clinicians' evaluation of leaks and the appearance of the pressure curve: a small pressure plateau is required and flow may be set accordingly) and rate will be started at 30 bpm (can be raised in steps of 5 bpm to max 50 bpm, according to PaCO2 levels).
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: NHFOV — Nasal high frequency oscillation ventilation (NHFOV) is used as the noninvasive supporting mode after extubation.
  Arms: NHFOV
Device: NCPAP — Nasal continuous positive airway pressure(NCPAP) is used as the noninvasive supporting mode after extubation.
  Arms: NCPAP
Device: NIPPV — Nasal intermittent positive pressure ventilation(NIPPV) is used as the noninvasive supporting mode after extubation.
  Arms: NIPPV

SUMMARY:
Respiratory distress syndrome (RDS) is the main cause of respiratory failure in preterm neonates, its incidence varying from 80% to 25% depending on gestational age.When optimal prenatal care is provided, the best approach to treat RDS, according to several recent trials,consists in providing continuous positive airway pressure (CPAP) from the first minutes of life using short binasal prongs or masks, followed by early selective surfactant administration for babies with worsening oxygenation and/or increasing work of breathing. Any effort should be done to minimize the time under invasive mechanical ventilation (IMV).Nonetheless, clinical trials have shown that a relevant proportion of preterm neonates fails this approach and eventually need IMV.The duration of IMV is a well known risk factor for the development of broncho-pulmonary dysplasia (BPD) - a condition associated with significant morbidity and mortality.

To minimize the duration of IMV, various non invasive respiratory support modalities are available in neonatal intensive care units (NICU). CPAP is presently the most common technique used in this regard. However, a systematic review has shown that non-invasive positive pressure ventilation (NIPPV) reduces the need for IMV (within one week from extubation) more effectively than NCPAP, although it is not clear if NIPPV may reduce need for intubation longterm and it seems to have no effect on BPD and mortality. NIPPV main drawback is the lack of synchronization, which is difficult to be accurately achieved and is usually unavailable. A more recent alternative technique is non-invasive high frequency oscillatory ventilation (NHFOV) which consists on the application of a bias flow generating a continuous distending positive pressure with oscillations superimposed on spontaneous tidal breathing with no need for synchronization. The physiological, biological and clinical details about NHFOV have been described elsewhere.

To date, there is only one small observational uncontrolled study about the use of NHFOV after extubation in preterm infants. Other relatively small case series or retrospective cohort studies suggested safety, feasibility and possible usefulness of NHFOV and have been reviewed elsewhere.The only randomized trial published so far compared NHFOV to biphasic CPAP,in babies failing CPAP and it has been criticized for methodological flaws and for not taking into account respiratory physiology.An European survey showed that, despite the absence of large randomized clinical trials, NHFOV is quite widely used, at least in some Countries and no major side effects are reported, although large data about NHFOV safety are lacking. This may be due to the relative NHFOV easiness of use but evidence-based and physiology-driven data are warranted about this technique.

DETAILED DESCRIPTION:
NHFOV should theoretically provide the advantages of invasive high frequency oscillatory ventilation (no need for synchronization, high efficiency in CO2 removal, less volume/barotrauma) and nasal CPAP (non-invasive interface, oxygenation improvement by the increase in functional residual capacity through alveolar recruitment). NHFOV should allow to increase mean airway pressure (Paw) avoiding gas trapping and hypercarbia, thanks to the superimposed high frequency oscillations. Therefore, NHFOV is more likely to be beneficial for those neonates requiring high distending pressure to open up their lungs, such as babies at high risk of extubation failure due to severity of their lung disease. This may also be the case of extremely preterm, BPD-developing neonates who have increased airway resistances, while they are subjected to a deranged alveolarization and lung growth. Neonates presenting with respiratory acidosis may also benefit from NHFOV. Several animal and bench studies investigated the physiology and peculiarities of NHFOV and these data should be used to conduct a physiology-guided trial in order to avoid errors done in the early trials about invasive high frequency ventilation.

This study will be the first large trial aiming to compare CPAP vs NIPPV vs NHFOV in preterm neonates after surfactant replacement and during their entire NICU stay, to reduce the total need of invasive ventilation. Since there is a lack of formal data regarding NHFOV safety, some safety outcomes will also be considered.Specific subgroup analysis will be conducted for pre-specified groups of patients who may most likely benefit from NHFOV, according to the above-described physiological characteristics.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 25+0 and 32+6 weeks;
* birth weight more than 600 g;
* supported with any type of endotracheal ventilation;
* Has not had first attempt at extubation(extubation readiness requires fulfilling of all the following criteria: a. Having received at least one loading dose of 20 mg/kg and 5 mg/kg daily maintenance dose of caffeine citrate; b. pH>7.20 PaCO2<=60 mmHg (these may be evaluated by arterialized capillary blood gas analysis or appropriately calibrated transcutaneous monitors. Venous blood gas values cannot be used); c. Paw <=7-8 cmH2O; d. FiO2<=0.30; e. sufficient spontaneous breathing effort, as per clinical evaluation).;
* Obtained parental consent. Informed consent will be obtained antenatally or upon neonatal intensive care unit admission.;

Exclusion Criteria:

* major congenital anomalies or chromosomal abnormalities;
* Presence of neuromuscular disease;
* Upper respiratory tract abnormalities; ;
* need for surgery known before the first extubation;
* Grade IV-intraventricular haemorrhage (IVH) occurring before the first extubation
* congenital lung diseases or malformations or pulmonary hypoplasia

Ages: 30 Minutes to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1493 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Every researchers can obtain the IPD after the study completely.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At Oct-22,2017,Suzhou,PR.China.

REFERENCES:
- [Derived] Zhu X, Li F, Shi Y, Feng Z, De Luca D; Nasal Oscillation Post-Extubation (NASONE) Study Group. Effectiveness of Nasal Continuous Positive Airway Pressure vs Nasal Intermittent Positive Pressure Ventilation vs Noninvasive High-Frequency Oscillatory Ventilation as Support After Extubation of Neonates Born Extremely Preterm or With More Severe Respiratory Failure: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2321644. doi: 10.1001/jamanetworkopen.2023.21644. PMID 37399009
- [Derived] Zhu X, Qi H, Feng Z, Shi Y, De Luca D; Nasal Oscillation Post-Extubation (NASONE) Study Group. Noninvasive High-Frequency Oscillatory Ventilation vs Nasal Continuous Positive Airway Pressure vs Nasal Intermittent Positive Pressure Ventilation as Postextubation Support for Preterm Neonates in China: A Randomized Clinical Trial. JAMA Pediatr. 2022 Jun 1;176(6):551-559. doi: 10.1001/jamapediatrics.2022.0710. PMID 35467744
- [Derived] Shi Y, De Luca D; NASal OscillatioN post-Extubation (NASONE) study group. Continuous positive airway pressure (CPAP) vs noninvasive positive pressure ventilation (NIPPV) vs noninvasive high frequency oscillation ventilation (NHFOV) as post-extubation support in preterm neonates: protocol for an assessor-blinded, multicenter, randomized controlled trial. BMC Pediatr. 2019 Jul 26;19(1):256. doi: 10.1186/s12887-019-1625-1. PMID 31349833

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2017 and May 2021, 1493 infants underwent randomization and data from 1440 were analyzed. A total of 53 infants were excluded from this analysis because missing data.
Pre-assignment Details: Between December 2017 and May 2021, 1493 infants underwent randomization and data from 1440 were analyzed. A total of 53 infants were excluded from this analysis because missing data.
Groups:
- NHFOV: neonates assigned to NHFOV will be started with the following boundaries:
  a) Paw of 10 cmH2O (can be changed in steps of 1 cmH2O within the range range 5- 16cmH2O); Paw will be titrated (within the range) according to open lung strategy, performing alveolar recruitment, similar to what is done in endotracheal high frequency oscillatory ventilation targeting a FiO2≤25-30%. Maximal allowed FiO2 will be 0.40 and SpO2 targets will be 90%-95%. b) frequency of 10Hz(can be changed in steps of 1Hz within the range 8-12Hz). c)Inspiratory time 50% (1:1).d)amplitude 25 cmH2O(can be changed in steps of 5 cmH2O within the range 25-50 cmH2o; amplitude will be titrated according to PaCO2.
  NHFOV: Nasal high frequency oscillation ventilation (NHFOV) is used as the noninvasive supporting mode after extubation.
Period: Overall Study
Arm/Group | NHFOV | NCPAP | NIPPV
Started | 497 | 501 | 495
Completed | 480 | 480 | 480
Not Completed | 17 | 21 | 15
Not completed — Lost to Follow-up | 17 | 21 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NHFOV | NCPAP | NIPPV | Total
Number analyzed (Participants) | 480 | 480 | 480 | 1440
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 29.4 (1.8) | 29.5 (1.7) | 29.4 (1.8) | 29.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296 | 208 | 292 | 796
  Male | 184 | 272 | 188 | 644
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Birth Weight [Mean (Standard Deviation); unit: g] | 1317 (353) | 1334 (366) | 1341 (318) | 1337 (352)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Invasive Mechanical Ventilation
Description: the total days of the baby supported with the ventilator
Time Frame: up to 8 weeks
Measure: Mean (Standard Deviation); unit: day
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
day | 6.3 (6.0) | 7.8 (7.2) | 7.3 (9.2)

2. Primary Outcome: Ventilator-free Days
Description: non-invasive ventilation was need after extubation
Time Frame: up to 8 weeks
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
day | 34 [17 to 52] | 32 [20 to 45] | 35 [21 to 52]

3. Primary Outcome: Number of Babies With Reintubation
Description: the total numbers of the baby supported with ventilator
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 63 | 123 | 84

4. Secondary Outcome: Number of Participants With Airleaks
Description: airleaks was diagnosed after extubation
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 4 | 3 | 9

5. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia(BPD)
Description: Bronchopulmonary dysplasia was defined, according to National Institutes of Health (NIH) criteria, by the receipt of any form of positive-airway-pressure support or a requirement for supplemental oxygen at 36 weeks. A requirement for supplemental oxygen at 36 weeks was defined as an FiO2 of 0.30 or more or
Time Frame: at gestational age of 36 weeks or at discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 163 | 184 | 182

6. Secondary Outcome: Number of Participants With Retinopathy of Prematurity> 2nd Stage
Description: Retinopathy of prematurity> 2nd stage was diagnosed after extubation
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 63 | 74 | 72

7. Secondary Outcome: Number of Participants With Neonatal Necrotizing Enterocolitis≥ 2nd Stage
Description: Neonatal necrotizing enterocolitis≥ 2nd stage was diagnosed after extubation
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 33 | 24 | 36

8. Secondary Outcome: Number of Participants With Intraventricular Hemorrhage>2nd Grade
Description: Intraventricular hemorrhage>2nd grade was diagnosed after extubation
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 48 | 63 | 59

9. Secondary Outcome: Number of Participants With Need for Postnatal Steroids
Description: steroids was used for chronic lung disease
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 63 | 77 | 98

10. Secondary Outcome: In-hospital Mortality
Description: the baby died in hospital
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 8 | 5 | 4

11. Secondary Outcome: Composite Mortality/BPD
Description: the baby was dead or diagnosed with BPD.
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 171 | 189 | 186

12. Secondary Outcome: Weekly Weight Gain
Description: Weekly weight gain (in grams/day) for the first 4 weeks of life or until NICU discharge, whichever comes first
Time Frame: during hospitalization for the first 4 weeks of life or until NICU discharge whichever came first, an average of 1 month
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
grams/day | 13.0 (5.3) | 12.1 (4.9) | 12.4 (6.4)

13. Secondary Outcome: Haemodynamically Significant Patent Ductus Arteriosus (PDA)
Description: hemodynamically significant patent ductus arteriosus (PDA), defined according to local NICU protocols
Time Frame: up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NHFOV | NCPAP | NIPPV
Number analyzed (Participants) | 480 | 480 | 480
Participants | 138 | 148 | 163

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Description: Nasal skin injury
Arm/Group | NHFOV | NCPAP | NIPPV
All-Cause Mortality (participants affected / at risk) | 8/480 | 5/480 | 4/480
Serious Adverse Events (participants affected / at risk) | 0/480 | 0/480 | 0/480
Other Adverse Events (participants affected / at risk) | 137/480 | 126/480 | 119/480
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NHFOV (N=480) | NCPAP (N=480) | NIPPV (N=480)
Nasal skin injury (Injury, poisoning and procedural complications) | 137 (137) | 126 | 119 (119)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03181958/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03181958/SAP_001.pdf
  • Informed Consent Form (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03181958/ICF_002.pdf